CLINICAL TRIAL: NCT01724632
Title: LIVE SMART: Smartphone Intervention for Weight Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, John Graham Thomas, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DK095779 (NIH)
Record Dates: First submitted 2012-11-06; First posted 2012-11-12 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group Treatment (Active Comparator): Participants who are assigned to group treatment will attend group meetings weekly for the first 6 months, then every 2 weeks for 6 months, and then monthly for the final 6 months. Participants will be weighed individually at the start of each group meeting.
  Interventions: Behavioral: Lifestyle Counseling
- Individual Treatment (Active Comparator): Participants who are assigned to individual treatment will attend one-on-one sessions with a weight loss counselor every month for 18 months.
  Interventions: Behavioral: Lifestyle Counseling
- Smartphone Treatment (Experimental): Participants who are assigned to smartphone treatment will use a smartphone to learn and practice weight loss skills. They will also attend one-on-one sessions with a weight loss counselor every month for 18 months.
  Interventions: Behavioral: Lifestyle Counseling

INTERVENTIONS:
Behavioral: Lifestyle Counseling — Participants receive instructions for making healthy changes to their diet and physical activity habits.

SUMMARY:
The purpose of this study is to compare three methods of delivering behavioral weight loss treatment.Participants are randomly assigned to one of three 18-month weight loss treatments (group, individual, or smartphone treatment). Participants who are assigned to group treatment will attend group meetings weekly for the first 6 months, then every 2 weeks for 6 months, and then monthly for the final 6 months. Participants who are assigned to individual treatment will attend one-on-one sessions with a weight loss counselor every month for 18 months. Participants who are assigned to smartphone treatment will use a smartphone to learn and practice weight loss skills. They will also attend one-on-one sessions with a weight loss counselor every month for 18 months. Assessment visits are conducted at baseline, 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (kg/m2) of 25-45.
* English language fluency
* Ability to read at a 6th grade level
* Availability to attend weekly treatment sessions in Providence, RI

Exclusion Criteria:

* Any heart condition that limits ability to participate in physical activity
* Chest Pain
* Any cognitive of physical limitation that would preclude use of a smartphone
* Serious mental illness
* Historical or current eating disorder
* Previous or planned bariatric surgery
* Use of weight loss medication
* Recent pregnancy or a plan to become pregnant in the next 6 months
* Participation in a study at the Weight Control and Diabetes Research Center within the last two years
* A weight loss of greater than 5% body weight in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2012-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Change from baseline to 18-months.

SECONDARY OUTCOMES:
Weight-related Behaviors | Change from baseline to 18-months.
  Questionnaire measures of diet, physical activity, and other weight related behaviors such as self-monitoring.

OTHER OUTCOMES:
Engagement with Smartphone Treatment system | Mueasured continuously for the 18-month treatment.
  Frequency and duration of use of intervention resources made available to the smartphone treatment arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Goldstein SP, Goldstein CM, Bond DS, Raynor HA, Wing RR, Thomas JG. Associations between self-monitoring and weight change in behavioral weight loss interventions. Health Psychol. 2019 Dec;38(12):1128-1136. doi: 10.1037/hea0000800. Epub 2019 Sep 26. PMID 31556659
- [Derived] Thomas JG, Bond DS, Raynor HA, Papandonatos GD, Wing RR. Comparison of Smartphone-Based Behavioral Obesity Treatment With Gold Standard Group Treatment and Control: A Randomized Trial. Obesity (Silver Spring). 2019 Apr;27(4):572-580. doi: 10.1002/oby.22410. Epub 2019 Feb 19. PMID 30779333
- [Derived] Bond DS, Thomas JG, O'Leary KC, Lipton RB, Peterlin BL, Roth J, Rathier L, Wing RR. Objectively measured physical activity in obese women with and without migraine. Cephalalgia. 2015 Sep;35(10):886-93. doi: 10.1177/0333102414562970. Epub 2014 Dec 4. PMID 25475207